CLINICAL TRIAL: NCT00343850
Title: Once Daily Versus Conventional Dosing of Asacol in the Maintenance of Quiescent Ulcerative Colitis: A Randomized Pilot Trial
Brief Title: Once Daily Versus Conventional Dosing of Asacol in the Maintenance of Quiescent Ulcerative Colitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Chicago (Other)
Collaborators: Procter and Gamble (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 14515A
Record Dates: First submitted 2006-06-21; First posted 2006-06-23 (Estimated); Last update posted 2013-01-10 (Estimated); Status verified 2013-01

CONDITIONS: Ulcerative Colitis
Keywords: idiopathic chronic inflammatory disease of large intestine; ulcerative colitis; inactive ulcerative colitis; chronic disease of large intestine; medication adherence; Asacol; mesalamine
MeSH Terms: conditions — Colitis, Ulcerative; Medication Adherence | interventions — Mesalamine

INTERVENTIONS:
Drug: Asacol (mesalamine)

SUMMARY:
The purpose of this study is to determine if taking Asacol once a day is as effective as taking Asacol twice or three times a day in keeping ulcerative colitis inactive, and to determine which dosing regimen is easiest to follow. Once daily dosing of Asacol is experimental, and has not been approved by the FDA. Dosing as three times daily is FDA approved.

This research is being done because the researchers want to learn what the best methods are for keeping ulcerative colitis inactive, and which way of taking Asacol is most helpful to subjects in continuing to take a medication to control their ulcerative colitis.

DETAILED DESCRIPTION:
Hypothesis: Asacol taken once a day is equally effective (non-inferior) as conventional (twice or three times a day) dosing at maintaining remission in quiescent ulcerative colitis.

Specific Aims:

1. To assess the efficacy of once daily Asacol in the short and long-term maintenance of remission in quiescent ulcerative colitis.
2. To assess the medication consumption rate (adherence) in patients prescribed once daily Asacol compared to a bid or tid regimen.

Background:

Ulcerative colitis (UC) is an idiopathic, chronic inflammatory disease of the large intestine characterized by episodes of relapse and remission. Relapses are often not predictable, although factors such as smoking cessation, chronic non-steroidal antiinflammatory use and psychological stress are thought to cause symptom exacerbation in some individuals.

Multiple studies have demonstrated the efficacy of aminosalicylates to induce and maintain remission in UC. Because of its chronic nature, therapy often must continue on an indefinite basis. Many patients openly admit they do not take their medications as prescribed; medication-taking probably makes patients more uncomfortably aware of their chronic illness status, they have a fear of long-term side effects from medications, and they question the need for medication in the setting of quiescent disease.

Previous work done at the University of Chicago demonstrated that using objective pharmacy data, rather than patient-derived information, the prevalence of medication non-adherence was 60% in patients with quiescent UC. The average amount of medication consumed was 70% of that prescribed. In a prospective study, those patients non-adherent with medications had a higher risk of relapse than those who consumed greater than 75% of their prescribed regimen.

It is difficult to get patients to take medication when they feel well, because the rationale for continued use remains unclear to them. The long-term goals of improving adherence are to reduce frequency of relapse, lower the incidence of long-term complications (i.e. colon cancer), and lower overall health costs. Making a regimen easy for patients is a key factor in increasing adherence.

Hussain recently showed that in normal subjects, median peak concentrations, trough concentrations and areas under the curve were similar for Asacol consumed either as a once or three times daily dosing regimen. Twenty-four hour urinary and fecal excretions, total recovery, and rectal tissue concentrations also were similar in both groups. The authors concluded that the steady-state pharmacokinetics of delayed-release Asacol was similar whether the drug was administered in three divided doses throughout the day or as a single daily dose.

There are data to suggest that the motility and function of the colon in patients with quiescent ulcerative colitis is similar to that of normal subjects. If this is indeed the case, then the pharmacokinetics of Asacol should mimic those of healthy controls. In a small pilot study, we were able to show that in a 6-month time, patients were no more likely to experience a flare of their disease and actually consumed more medication in a once daily regimen than in a standard regimen. The aim of this study is to test this hypothesis in a larger number of patients, and assess the efficacy of once daily Asacol in patients with quiescent ulcerative colitis compared to a twice or three times daily regimen. In addition, we wish to compare the rates of medication consumption between groups over a prolonged period of time.

Methods:

Patients eligible will be asked to sign informed consent prior to participation. As part of the consent process, the phone number of the patient pharmacy will be collected. Patients will then be randomized to one of two groups: once daily or usual (twice daily or three times daily) therapy. Assignment will be via the use of opaque sealed envelopes, containing assignment based on a randomization table. Once enrolled, each patient will be assigned a study number, which will be used on the questionnaires to maintain confidentiality. The patients will be instructed to conceal their regimen from any research investigator.

Patients will be followed prospectively and assessed at 3 month intervals from enrollment. The three and nine-month follow up will be via phone contact by one of the study nurses. Disease assessment and quality of life will be obtained by the nurse in a standard fashion. At time intervals 6 and 12 months, patients will be assessed during a scheduled clinic visit, using the same assessment tools along with a physical exam. These visits will not be additional or extra visits, but part of standard of care for ulcerative colitis. There will be no additional blood draws or endoscopy as part of the protocol, lab work and endoscopy for patient care as determined by each treating physician will be documented.

Medication consumption rates at months 3, 6, 9 and 12 will be calculated using pharmacy data as obtained by telephone by the PI and the validated formula as described by Steiner and colleagues. The end point of the study is disease relapse or the 12-month study period. An investigator blinded to the treatment regimen will assess the outcomes and medication consumption rates for each group. Patients experiencing a flare during the study period will be treated as deemed necessary by their treating physician.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients over the age of 18 followed at the University of Chicago Outpatient Gastroenterology Clinic will be eligible. Patients must have documentation of ulcerative colitis by standard criteria, and be in remission for at least 4 months prior to study entry. Remission for this study will be defined clinically, as the absence of all of the following: blood in the stools, urgency, or cramping. Patients must be taking a regimen of Asacol (Asacol, Procter and Gamble, Cincinnati Ohio) for maintenance of quiescent disease

Exclusion Criteria:

* Exclusion criteria include documented disease activity in the past four months, hospitalization or steroid use for disease activity in the previous 4 months, or the use of other immunomodulators to induce remission. Patients with a history of other diarrheal illnesses such as diarrhea-predominant Irritable Bowel Syndrome, C difficile colitis, use of known diarrheal drugs will also be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2006-09; Primary Completion 2007-03 (Actual); Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
calculation of medication consumption rates at months 3, 6, 9 and 12
disease relapse
12-month study period

CONTACTS AND LOCATIONS:
Overall Officials: Sunanda Kane, MD, Principal Investigator — University of Chicago
Locations (1):
- The University of Chicago, Chicago, Illinois, United States

REFERENCES:
- [Background] Silverstein MD, Lashner BA, Hanauer SB. Cigarette smoking and ulcerative colitis: a case-control study. Mayo Clin Proc. 1994 May;69(5):425-9. doi: 10.1016/s0025-6196(12)61637-1. PMID 8170192
- [Background] Fraga XF, Vergara M, Medina C, Casellas F, Bermejo B, Malagelada JR. Effects of smoking on the presentation and clinical course of inflammatory bowel disease. Eur J Gastroenterol Hepatol. 1997 Jul;9(7):683-7. doi: 10.1097/00042737-199707000-00007. PMID 9262977